CLINICAL TRIAL: NCT03328026
Title: A Phase I/II Study of the SV-BR-1-GM Regimen in Metastatic or Locally Recurrent Breast Cancer Patients in Combination With Retifanlimab
Brief Title: Combination Study of SV-BR-1-GM With Retifanlimab
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BriaCell Therapeutics Corporation (Industry)
Collaborators: LumaBridge (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI-ROL-001
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Breast Neoplasm; Metastatic Breast Cancer; Breast Cancer Metastatic
Keywords: Breast Cancer; Metastatic Breast Cancer; MBC; Immunotherapy; Cancer Vaccine
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SV-BR-1-GM, retifanlimab combination original sequence (Experimental): Subjects will be treated with the SV-BR-1-GM regimen in combination with retifanlimab with cycles every 3 weeks
  Interventions: Biological: SV-BR-1-GM; Drug: Low dose cyclophosphamide; Drug: Interferon Inoculation; Drug: retifanlimab
- SV-BR-1-GM, retifanlimab combination alternative sequence (Experimental): Subjects will be treated with the SV-BR-1-GM regimen in combination with retifanlimab as follows:
  Cycle 1: SV-BR-1-GM only Cycle 2: resume retifanlimab on Day 2±1 Cycle 3 and beyond: retifanlimab can be administered on Day -2, Day 0, 1, 2, or 3.
  Interventions: Biological: SV-BR-1-GM; Drug: Low dose cyclophosphamide; Drug: Interferon Inoculation; Drug: retifanlimab

INTERVENTIONS:
Biological: SV-BR-1-GM — SV-BR-1-GM inoculation intradermally at 4 sites.
Drug: Low dose cyclophosphamide — Pretreatment with low dose cyclophosphamide 2-3 days prior to SV-BR-1-GM inoculation.
  Other Names: Cytoxan
Drug: Interferon Inoculation — Post-inoculation low dose Interferon into the vaccination sites ~2 days after SV-BR-1-GM inoculation.
Drug: retifanlimab — retifanlimab 375mg administered as an intravenous infusion over 30-60 minutes every 3 weeks per randomization
  Other Names: INCMGA00012

SUMMARY:
This is an open-label, phase I/II double arm study of the SV-BR-1-GM regimen in combination with retifanlimab in patients with metastatic or locally recurrent breast cancer who have failed standard therapy.

Patients will receive the SV-BR-1-GM regimen with combination immunotherapy. There will be an initial evaluation of the combination of the SV-BR-1-GM regimen with retifanlimab every 3 weeks. If this is found to be safe and well tolerated in a cohort of at least 12 patients (dose-limiting toxicities (DLTs) in less than 30% of the patients evaluated), then an expansion cohort of up to 24 patients will be treated with that combination. These will be randomized to two regimens differing in the timing of checkpoint inhibitor administration.

DETAILED DESCRIPTION:
This is an open-label, phase I/II double arm study of the SV-BR-1-GM regimen in combination with retifanlimab in patients with metastatic or locally recurrent breast cancer who have failed standard therapy.

Patients will receive the SV-BR-1-GM regimen with combination immunotherapy. There will be an initial evaluation of the combination of the SV-BR-1-GM regimen with retifanlimab every 3 weeks. If this is found to be safe and well tolerated in a cohort of at least 12 patients (dose-limiting toxicities (DLTs) in less than 30% of the patients evaluated), then an expansion cohort of up to 24 patients will be treated with that combination. These will be randomized to two regimens differing in the timing of retifanlimab administration as noted below.

The SV-BR-1-GM regimen consists of:

* Pre- SV-BR-1-GM cyclophosphamide 2-3 days prior to SV-BR-1-GM inoculation
* SV-BR-1-GM inoculation on day 0
* Interferon - at the inoculation sites 2 (±1) day post-SV-BR-1-GM

Combination therapy with retifanlimab (anti-PD-1) will be given per one of two randomized treatment arms as follows:

The SV-BR-1-GM regimen with retifanlimab will be administered every 3 weeks (± 3 days), except when approved by the Investigator in consultation with the Medical Monitor. Note that hormonal therapy (e.g., aromatase inhibitors) is permitted if ongoing, but may be added while the patient is on this study only with the Medical Monitor's approval (e.g. for hormone receptor positive patients who are deriving clinical benefit but have not achieved a CR after >6 cycles of therapy).

Following the initial cohort, an expansion cohort of 24 patients will be randomized 1:1 into two arms with differences in initial treatment sequences: original sequence and alternative sequence. The original sequence arm will receive treatment in the same schedule as the initial cohort. Subjects in the alternative sequence will skip retifanlimab in Cycle 1, and resume retifanlimab on Day 2±1 at Cycle 2. Starting Cycle 3, retifanlimab can be administered either on Day -2/-3, Day 0 or Day 2±1. Patients will be screened to ensure they fulfill the enrollment criteria. Screening must be performed within 30 days of initiating therapy. Imaging studies must be performed within 30 days of initiating therapy for the initial 12 patients, and within 14 days for the expansion cohort (randomized portion), unless approved by the Sponsor. For subjects in expansion cohort participating in the substudy, the CD8 attenuation CT scan cannot be used for the baseline image. However, patients can be immediately scanned after the low dose attenuation scan. In the expansion cohort randomized portion of the trial, imaging must be performed within 14 days of the start of study treatment. Patients will be evaluated every 3 weeks during the study, including all safety assessments. Imaging studies will be performed every 8-12 weeks during study participation.

Pharmacodynamic assessments, including evaluation of the immune response to SV-BR-1-GM will also be performed during screening visit (substudy only), during Cycle 1, every 8-12 weeks and End of Treatment. Subsequent periodic assessments will be every 8-12 weeks from the first periodic assessment. Patients who develop progressive disease may remain on treatment for up to 6 weeks to obtain a confirmatory scan per iRECIST; or as long as the Investigator feels they are deriving clinical benefit with Medical Monitor approval. For patients who come off treatment, a final assessment will be carried out 2-4 weeks following the last dose of SV-BR-1-GM, including all safety assessments. Off-treatment subjects will continue to be followed for survival analysis every 3 months (e.g., by phone call) for at least 5 years or until death.

For the CD8 ImmunoPET sub-study, ten (10) patients will be recruited from select invited sites only, and will undergo CD8 ImmunoPET evaluation at baseline and following 3 cycles of SV-BR-1-GM therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Have histological confirmation of breast cancer with recurrent and/or metastatic lesions, as per the investigational site, and have failed prior therapy.
2. Patients with persistent disease and local recurrence must not be amenable to local treatment.
3. For patients with metastatic disease:

   1. Human epidermal growth factor 2 (HER2) positive and estrogen receptor (ER) or progesterone receptor (PR) positive tumors: must be refractory to hormonal therapy (e.g., aromatase inhibitor, tamoxifen or fluvestrant) and previously treated with at least 2 regimens including at least two anti-HER2 agents (e.g., trastuzumab and pertuzumab).
   2. HER2 negative and either ER or PR positive tumors: must be refractory to hormonal therapy (e.g. aromatase inhibitor, tamoxifen or fluvestrant) and previously treated with at least 2 chemotherapy containing regimens. (e.g. CDK4/6 inhibitor, PIK3CA inhibitor, etc)
   3. HER2 positive and ER and PR negative tumors: must have failed at least 2 regimens including at least two anti-HER2 agents (e.g., trastuzumab and pertuzumab).
   4. Triple Negative tumors: Must have exhausted other available therapies including prior treatment with a taxane and carboplatin.

   Patients with new or progressive breast cancer metastatic to the brain will be eligible provided:
   1. The brain metastases must be clinically stable (without evidence of progressive disease by imaging) for at least 4 weeks prior to first dose
   2. Must have received prior radiation therapy for brain metastases or be ineligible for radiation therapy
   3. There is no need for steroids and patients have not had steroids for at least 2 weeks
   4. No individual tumor size is >50 mm
   5. Tumor is not impinging on Middle Cerebral Artery/speech-motor strip
   6. If surgically debulked, must be healed from surgery and at least 3 weeks have elapsed since general anesthesia
   7. Patients consent to MRI studies at 3-4 week intervals until evidence of tumor regression on at least 2 imaging studies. In no case, will the interval between MRI studies be longer than 3 months. MRI studies may be introduced at any time should the patients develop new or clearly worsening symptoms and/or introduction of steroids
4. Be 18 years of age or older and female
5. Have expected survival of at least 4 months
6. Have adequate performance status (ECOG 0-1) Patients with ECOG of 2 may be admitted only with Sponsor approval.
7. Have provided written informed consent

Exclusion Criteria:

1. Concurrent or recent chemotherapy, immunotherapy (except the SV-BR-1-GM regimen), or general anesthesia/major surgery within 21 days. Patients must have recovered from all known or expected toxicities from previous systemic treatment and passed a treatment-free "washout" period of 3 weeks before starting this program (8 weeks for patients receiving nitrosourea or mitomycin). Prior immune related toxicity should not have exceeded Grade 2 (with exception of endocrinopathy).
2. Radiotherapy within 14 days of first dose of study treatment with the following caveats:

   1. 28 days for pelvic radiotherapy.
   2. 8 weeks for brain metastases
   3. 6 months for thoracic region radiotherapy that is > 30 Gy in 2 Gy fractions.
3. Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline (with the exception of any grade of alopecia and anemia not requiring transfusion support). Endocrinopathy, if well-managed, is not exclusionary and should be discussed with medical monitor.
4. Participant has not recovered adequately from toxicities and/or complications from surgical intervention before starting study drug.
5. History of clinical hypersensitivity to the designated combination immunotherapy, GM-CSF, Interferon, yeast, beef, or to any components used in the preparation of SV-BR-1-GM.
6. History of clinical hypersensitivity to any of the immunotherapies proposed for combination treatment or their excipients.
7. Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (e.g., antihistamines and corticosteroids) or known allergy or hypersensitivity to any component of retifanlimab or formulation components.
8. Serum creatinine OR Measured or calculated Creatinine Clearance (CrCl) (GFR can also be used in place of creatinine or CrCl) >1.5 × ULN OR <30 mL/min for participants with creatinine levels >1.5 × institutional ULN.
9. Absolute granulocyte count <1000; platelets <100,000; hemoglobin ≤ 8 g/L.
10. Bilirubin ≥ 1.5 × ULN unless conjugated bilirubin ≤ ULN; alkaline phosphatase >5x upper limit of normal (ULN); ALT/AST >2x ULN. For patients with hepatic metastases, ALT/AST >5x ULN is exclusionary.
11. INR or PT or aPTT > 1.5 × ULN, unless the participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants. Note: See the restricted medications list in protocol section 5.9. If an alternative cannot be found, the participant cannot be enrolled.
12. Receiving any medication listed in the prohibited medication (section 5.10 of the protocol).
13. Proteinuria >1+ on urinalysis or >1 gm/24hr.
14. History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful. Screening corrected QT interval (QTc) interval >480 milliseconds is excluded (corrected by Fridericia or Bazett formula). In the event that a single QTc is >480 milliseconds, the participant may enroll if the average QTc for the 3 ECGs is <480 milliseconds.

16. Left ventricular ejection fraction (LVEF as determined by cardiac echo or MUGA scan) below the normal limits of the institutions' specific testing range.

17. New York Heart Association stage 3 or 4 cardiac disease. 18. A pericardial effusion of moderate severity or worse. 19. Symptomatic pleural effusion or ascites. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.

20. Any woman of childbearing potential (i.e., has had a menstrual cycle within the past year and has not been surgically sterilized), unless she: agrees to take appropriate precautions to avoid becoming pregnant during the study (with at least 99% certainty, see Appendix A for permitted methods) and has a negative serum pregnancy test within 7 days prior to starting treatment.

21. Men must have been sterile or, if they were potentially fertile/reproductively competent, should take appropriate precautions to avoid fathering a child for the duration of the study.

22. Women who are pregnant or nursing. 23. Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 3 years of study entry with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the participant has been disease-free for > 1 year, after treatment with curative intent.

24. Patients who are HIV positive (by self-report) and have clinical or laboratory features indicative of AIDS.

25. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.

25. Has had an allogeneic tissue/solid organ transplant. 26. Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.

27. Patients with a history of colitis. 28. Has a history of (non-infectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease.

29. Known active HBA, HBV, or HCV infection, as defined by elevated transaminases with the following serology: positivity for HAV IgM antibody, anti-HCV, anti-HBc IgG or IgM, or HBsAg (in the absence of prior immunization).

30. Active infections requiring systemic therapy.

a. All antibiotic therapy within 28 days of initiating treatment must be recorded 31. Has a known history of active tuberculosis (TB; Bacillus tuberculosis). 32. Patients with severe psychiatric (e.g., schizophrenia, bipolar, or borderline personality disorder) or other clinically progressive major medical problems, unless approved by the Investigator in consultation with the medical monitor.

33. Has received a live vaccine within 28 days of the planned start of study drug. Note: examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live-attenuated vaccines and are not allowed.

34. Patients may not be on a concurrent clinical trial, unless approved by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Adverse Events (AEs), including Serious Adverse Events (SAEs), that occur in patients treated with SV-BR-1-GM administered in combination with INCMGA00012 (retifanlimab) [Safety] | Through study completion, an average of 1 year
  To evaluate the safety of SV-BR-1-GM as assessed by:
  o Adverse Events (AEs), including Serious Adverse Events (SAEs)
Evaluate the Proportion of Patients with Abnormalities in Safety Laboratory Parameters that occur in patients treated with SV-BR-1-GM administered in combination with INCMGA00012 (retifanlimab) [Safety] | Through study completion, an average of 1 year
  To evaluate the safety of SV-BR-1-GM as assessed by:
  o The Proportion of Patients with Abnormalities in Safety Laboratory Parameters
Evaluate changes in the electrocardiogram QT interval that occur in patients treated with SV-BR-1-GM administered in combination with INCMGA00012 (retifanlimab)[Safety] | Through study completion, an average of 1 year
  To evaluate the safety of SV-BR-1-GM as assessed by:
  o Electrocardiograms (ECG) with measurement of the QT interval

SECONDARY OUTCOMES:
Evaluate the tumor response to SV-BR-1-GM (ORR) when administered in combination with INCMGA00012 (retifanlimab) | Through study completion, an average of 1 year
  Tumor response as assessed by:
  o Objective response rate (ORR), defined as complete response (CR) or partial response (PR) per RECIST 1.1
Evaluate the tumor response to SV-BR-1-GM (Non-progression) when administered in combination with INCMGA00012 (retifanlimab) | Through study completion, an average of 1 year
  Tumor response as assessed by:
  o Non-progressive rate, defined as CR, PR or stable disease (SD) per iRECIST
Evaluate the tumor response to SV-BR-1-GM (Durability) when administered in combination with INCMGA00012 (retifanlimab) | Through study completion, an average of 1 year
  Tumor response as assessed by:
  o Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, FACS, Study Director — LumaBridge LLC
Locations (14):
- United States (14):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami/Sylvester at Plantation, Plantation, Florida
  - Carle Cancer Institute, Urbana, Illinois
  - Cancer Center of Kansas (CCK), Wichita, Kansas
  - The Center for Cancer and Blood Disorders a division of American Oncology Partners MD, Bethesda, Maryland
  - St Vincent-Frontier Cancer Center, Billings, Montana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Overlook Medical Center Oncology Research, Atlantic Health System, Summit, New Jersey
  - Manhattan Hematology Oncology Associates (MHOA), Manhattan, New York
  - Mary Crowley Cancer Research, Dallas, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Hematology-Oncology Associates of Fredericksburg, Inc, Fredericksburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://briacell.com/
- See also: CRO Website — http://www.lumabridge.com/